CLINICAL TRIAL: NCT02372981
Title: Doppler-guided Haemorrhoidal Artery Ligation With Suture Mucopexy vs. Suture Mucopexy Alone for the Treatment of Grade III Haemorrhoids: A Prospective-randomised Controlled Trial
Brief Title: Doppler-guided Haemorrhoidal Artery Ligation With Suture Mucopexy vs. Suture Mucopexy Alone
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University Innsbruck (Other)
Responsible Party: Principal Investigator, Felix Aigner, ao. Univ.-Prof. Dr. med., Medical University Innsbruck
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MUI
Record Dates: First submitted 2015-02-06; First posted 2015-02-26 (Estimated); Last update posted 2015-02-26 (Estimated); Status verified 2015-02

CONDITIONS: Third Degree Hemorrhoids

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- DG-HAL with mucopexy (Experimental): Mucopexy with DG-HAL is performed using a specific device consisting of a proctoscope equipped with a Doppler probe and a light source. The proctoscope model in our study has a sliding part comprising the operating window and Doppler probe for better proximal and distal movement without repositioning the proctoscope during mucopexy.
  Interventions: Device: mucopexy +/- Doppler-guided haemorrhoidal artery ligation
- mucopexy alone (Active Comparator): Mucopexy without DG-HAL is performed using the same specific device consisting of a proctoscope equipped with a Doppler probe and a light source as described above.
  Interventions: Device: mucopexy +/- Doppler-guided haemorrhoidal artery ligation

INTERVENTIONS:
Device: mucopexy +/- Doppler-guided haemorrhoidal artery ligation — Mucopexy with or without DG-HAL is performed using a specific device consisting of a proctoscope equipped with a Doppler probe and a light source. The proctoscope model in our study has a sliding part comprising the operating window and Doppler probe for better proximal and distal movement without repositioning the proctoscope during mucopexy.

SUMMARY:
Novel minimally invasive techniques were established for prolapsing haemorrhoids to minimise the drawbacks of the golden standard of haemorrhoidal treatment, conventional haemorrhoidectomy techniques. Ligation techniques, such as Doppler-guided haemorrhoidal artery ligation (DG-HAL), were introduced to reduce the arterial inflow of the AVP and thus prevent the haemorrhoidal zone from being part of the continence system. Apart from inappropriate application of this surgical alternative for higher grade haemorrhoids, high recurrence rates of up to 38% after DG-HAL are due to technical failure of the ligation technique itself. This is a prospective randomised controlled trial to evaluate the efficacy of additional Doppler-guided ligation of submucosal haemorrhoidal arteries in patients with symptomatic grade III haemorrhoids.

DETAILED DESCRIPTION:
All consecutive patients with symptomatic grade III haemorrhoids are randomly allocated to one of the two study arms: (A) DG-HAL with mucopexy or (B) mucopexy alone. Endpoints are pain, faecal incontinence, bleeding, residual prolapse and vascularisation of the anorectal vascular plexus. Vascularisation of the anorectal vascular plexus is assessed by transperineal contrast enhanced ultrasound.

ELIGIBILITY:
Inclusion Criteria:

* grade III haemorrhoids
* ≥18 years of age

Exclusion Criteria:

* malignant gastrointestinal disease
* inflammatory bowel disease
* any type of proctological intervention (i.e., fistula surgery)
* recurrent haemorrhoidal disease
* anorectal trauma in the history

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2010-10; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
pain assessment wit 1-month-pain diary | 1 month

REFERENCES:
- [Derived] Aigner F, Kronberger I, Oberwalder M, Loizides A, Ulmer H, Gruber L, Pratschke J, Peer S, Gruber H. Doppler-guided haemorrhoidal artery ligation with suture mucopexy compared with suture mucopexy alone for the treatment of Grade III haemorrhoids: a prospective randomized controlled trial. Colorectal Dis. 2016 Jul;18(7):710-6. doi: 10.1111/codi.13280. PMID 26787597